CLINICAL TRIAL: NCT05039788
Title: Monocentric Observational Study to Determine the Relationship Between Arterial Hypertension and Hypervolaemia, Defined by Self-measurement of Impedancemetry in Kidney Transplant Recipients Under 6 Months Old
Brief Title: Observational Single-center Study of the Relationship Between Arterial Hypertension and Hypervolemia Defined by Self-measurement of Impedancemetry in Kidney Transplant Patients With Transplantation Less Than 6 Months Old
Acronym: HTAôConnect
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC20_0484
Record Dates: First submitted 2021-06-08; First posted 2021-09-10 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Kidney Transplant Patients
Keywords: Hypertension; Hypervolemia; Self-measurement; Connected
MeSH Terms: conditions — Hypertension; Edema | interventions — Blood Pressure; Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Measurement of systolic and diastolic blood pressure, impedancemetry, weight, creatinemia and Pro-BNP measurements — Measurement of systolic and diastolic blood pressure, impedancemetry, weight, creatinemia and Pro-BNP measurements At D30 and D90
  Measurement of systolic and diastolic blood pressure, impedancemetry, weight, 3 times a week between D30 and D90 post-transplant,

SUMMARY:
The working hypothesis is that hypertension during the first post-transplant trimester is partly explained by the patient's hypervolemia. The main objective of the single-center observational study "HTA ô Connect" is to study the relationship between hypertension and extracellular hyperhydration, thanks to repeated self-measurements of blood pressure and impedancemetry between the 30th and the 90th day post-transplant, in 150 incident kidney transplant patients from our department, the ITUN (Institute of Urology-Nephrology Transplantation).

The study population involves 150 incident kidney transplant patients, presenting to the Nantes University Hospital Transplant Institute for 1 month (D30), and presenting with hypertension ≥ 140/90mmHg and not treated with a diuretic.

Data collected at the patients' homes will be used to establish a relationship between blood pressure and extracellular water volume. The data collected will not be used to follow up patients who participated in the study in this first stage of exploration.

DETAILED DESCRIPTION:
Evaluation parameters

1. Blood pressure :

   * At inclusion and at the end of the study (in consultation at D30 and D90, respectively), blood pressure will be measured 3 times after a few minutes of rest in a sitting position Hypertension in consultation will be defined by values > 140/90 mmHg.
   * Between D30 and D90, blood pressure will be measured by self-measurement using DM-certified devices, 3 times in the morning at breakfast and in the evening before bedtime, in a sitting position after a few minutes of rest. The operation will be repeated 3 days a week (Monday to Wednesday) between the 30th and the 90th day post-transplant. Self-measurement hypertension will be defined by values > 135/85 mmHg. Self-measurement blood pressure data will be directly transmitted to the "INTEGRALIS" specialty medical record of transplant patients at the ITUN via the epatient application (https://www.idbc.fr/e-patient/).
2. Weight :

   * Weight will be measured only once at the inclusion consultation (D30) and at the end of the study (D90).
   * Between D30 and D90 the weight will be measured by self-measurement using DM certified scales. The operation will be repeated once in the morning and once in the evening at the time of blood pressure measurements, 3 days a week (Monday to Wednesday) between the 30th and the 90th day after transplantation. The data from the self-measurement of weight will be directly transmitted to the "INTEGRALIS" medical record of the transplanted patients at the ITUN
3. Impedance measurement :

   * At inclusion and at the end of the study in consultation, respectively at D 30 and D90, impedancemetry will be measured once
   * Between D30 and D90, impedancemetry measurements will be collected at the same time as blood pressure measurements at the patients' homes by self-measurement 3 times in the morning and 3 times in the evening, 3 days a week (from Monday to Wednesday) between the 30th and the 90th day after transplantation. The impedancemetry will be collected with the help of a bluetooth-connected BIODYLIFEZM self-measurement device. The impedancemetry data collected via bluetooth will be directly transmitted to the "INTEGRALIS" specialty medical record of the transplanted patients at the ITUN.

ELIGIBILITY:
Inclusion Criteria :

* Age ≥ 18 years
* Blood pressure ≥ 140/90mmHg on 3 occasions and according to the recommendations of the French Society of Hypertension (6) at the M1 consultation
* Isolated kidney transplant patient
* BMI between 16 and 34 kg/cm2
* Not opposed to the research

Exclusion Criteria :

* History of non-renal transplantation
* Patients treated with diuretics on the day of inclusion
* Minors, adults under guardianship and protected persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population involves 150 incident kidney transplant patients, presenting to the Nantes University Hospital Transplant Institute for 1 month (D30), and presenting with hypertension ≥ 140/90mmHg recorded in the outpatient clinic at the Nantes University Hospital, according to the recommendations of the French Society of Arterial Hypertension (6) and not treated with a diuretic.
  There will be no emergency inclusion. Recently transplanted patients will come regularly, between 1 and 2 times per week, to the Nantes University Hospital during the first month. The study will be presented to them during this period and they will be included at the D30 (M1) consultation.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-10-14 (Actual); Primary Completion 2025-10-14 (Estimated); Study Completion 2025-12-14 (Estimated)

PRIMARY OUTCOMES:
Correlation between Hypertension and extracellular hyperhydration | Day 90
  Hypertension will be assessed by measurement of blood pressure
Correlation between Hypertension and extracellular hyperhydration | Day 90
  Extracellular hyperhydration will be measured by impedance measurement

SECONDARY OUTCOMES:
hypertension measurement | For 3 month post-transplant
  Blood pressure :
  At inclusion and at the end of the study (in consultation at Day 30 and Day 90, respectively), blood pressure will be measured 3 times after a few minutes of rest in a sitting position Hypertension in consultation will be defined by values > 140/90 mmHg.
  • Between Day 30 and D90, blood pressure will be measured by self-measurement using DM-certified devices, 3 times in the morning at breakfast and in the evening before bedtime, in a sitting position after a few minutes of rest. The operation will be repeated 3 days a week (Monday to Wednesday) between the 30th and the 90th day post-transplant. Self-measurement hypertension will be defined by values > 135/85 mmHg.
Impedance measurement | For 3 month post-transplant
  At inclusion and at the end of the study in consultation, respectively at Day 30 and D90, impedancemetry will be measured once.
  • Between Day 30 and Day 90, impedancemetry measurements will be collected at the same time as blood pressure measurements at the patients' homes by self-measurement 3 times in the morning and 3 times in the evening, 3 days a week (from Monday to Wednesday) between the 30th and the 90th day after transplantation.
Weight measurement | day 30
  Weight will be measured only once at the inclusion consultation
Weight measurement | Day 90
  Weight will be measured at the end of the study .
Weight measurement | 3 days a week between the 30th and the 90th day after transplantation.
  The weight will be measured by self-measurement using DM certified scales.
Correlation between repeated systolic and diastolic blood pressure self-measurements and patient weight | Day 90
  blood pressure will be measured 3 times after a few minutes of rest in a sitting position Hypertension in consultation will be defined by values > 140/90 mmHg.
  * Between Day 30 and D90, blood pressure will be measured by self-measurement using DM-certified devices, 3 times a week.
  * Weight will be measured only once at the inclusion consultation (Day30) and at the end of the study (Day 90).
  * Between Day30 and Day 90 the weight will be measured by self-measurement using DM certified scales.
Correlation between repeated self-measurements of extracellular hyperhydration | 3 times a week
  Impedance measurement
Correlation between repeated self-measurements of extracellular hyperhydration | 3 times a week
  Weight
Correlation between repeated self-measurement of systolic and diastolic blood pressure and creatinemia and pro-BNP blood | Day 90
  Composites criteria :
  Systolic and diastolic blood pressure will be assessed by measurement of blood pressure Plasma creatinine and proBNP will mesuread by a blood test
Correlation between repeated self-measurement of extracellular hyperhydration indices by impedancemetry and creatinemia and pro-BNP blood | Day 90
  Composites criteria :
  Extracellular hyperhydration will be measured by impedance measurement Plasma creatinine and proBNP will mesuread by a blood test

CONTACTS AND LOCATIONS:
Overall Officials: Claire GARANDEAU, PH, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: No